CLINICAL TRIAL: NCT06300606
Title: Is the Regional Anesthesia Technique Painful? an Evaluation Using the Nociception Index Level (NOL), a New Pain Monitoring, and Algiscore, a Multidimensional Pain Score
Brief Title: Nociception Index Level (NOL) Perioperative Monitoring During Regional Anesthesia
Acronym: NOL and LRA
Status: Recruiting | Type: Observational
Sponsor: American Hospital of Paris (Other)
Collaborators: Nataliya KARASHCHUK (Unknown); Briana LUI (Unknown); Thierry GUENOUN (Unknown); Stephane ROMANO (Unknown)
Responsible Party: Principal Investigator, Gilles BOCCARA, anesthesiologist, MD, PhD, American Hospital of Paris
Other Study IDs: NOL1 and RA
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Regional Anesthesia; Pain; Intraoperative Monitoring
Keywords: nociception; regional anesthesia; intraoperative monitoring; NOL monitor
MeSH Terms: conditions — Pain | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NOL monitoring — Prospective observational study to assess pain during regional anesthesia for upper limb orthopedic surgery using NOL monitoring and the Algoplus pain scale
  Other Names: regional anesthesia

SUMMARY:
This prospective observational study was conducted to assess pain using NOL index under locoregional anesthesia for orthopedic surgery of the upper limb. We included 50 consecutive adult patients scheduled for orthopedic surgery of the upper limb under locoregional anesthesia. The locoregional anesthesia was performed under ultrasound, with or without neurostimulation. Intraoperative pain is assessed using NOL index monitoring, ALGISCORE and Numerical Scale, and second point study is the midazolam and propofol requirement.

DETAILED DESCRIPTION:
Introduction: Intraoperative pain assessment is difficult and based on indirect parameters of sympathetic-parasympathetic system stimulation. Recently, the Nociception Level index (NOL™) providing a value from combination of multiple physiological parameters to measure pain has been developed to enable intraoperative pain monitoring during general anesthesia. While this monitoring has also been used postoperatively in awake patients, data are scarce to assess pain under locoregional anesthesia. This study was conducted to assess pain using NOL index under locoregional anesthesia for orthopedic surgery of the upper limb.

Method: 50 consecutive patients scheduled for orthopedic surgery of the upper limb under locoregional anesthesia were included. Exclusion criteria were emergencies, request for general anesthesia, and patients under 18 years of age. All patients were informed and consented to the technique of locoregional anesthesia and pain monitoring without change of practice. After premedication with oral hydroxyzine, locoregional anesthesia was performed under ultrasound, with or without neurostimulation. Monitoring began as soon as the venous infusion was started, and parameters were recorded at the time of locoregional anesthesia, tourniquet inflation, surgical incision, skin closure and dressing.

Pain is also assessed using the ALGISCORE by the nurse and the numerical scale (0 to 5) and satisfaction score at the end of the procedure. The need to administer midazolam or propofol at the anesthetist's discretion is noted, as is the effectiveness of locoregional anesthesia (conversion to general anesthesia). Data were analyzed using Friedman and Mann-Whitney tests.

ELIGIBILITY:
Inclusion Criteria:

scheduled upper limb orthopedic surgery under regional anesthesia

Exclusion Criteria:

Patient less than 18 years old emergency surgery patient refusal of regional anesthesia chronic neurocognitive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all the patients scheduled to undergo an upper limb orthopedic surgery under regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
pain score | intraoperative
  Nociception index level monitoring NOL
pain score | intraoperative
  ALGOPLUS pain scale

SECONDARY OUTCOMES:
sedative requirement | intraoperative
  propofol
anxiolytic requirement | intraoperative
  midazolam
failure of regional anesthesia | intraoperative
  general conversion or sufentanil requirement

CONTACTS AND LOCATIONS:
Locations (1):
- Gilles BOCCARA, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijer FS, Niesters M, van Velzen M, Martini CH, Olofsen E, Edry R, Sessler DI, van Dorp ELA, Dahan A, Boon M. Does nociception monitor-guided anesthesia affect opioid consumption? A systematic review of randomized controlled trials. J Clin Monit Comput. 2020 Aug;34(4):629-641. doi: 10.1007/s10877-019-00362-4. Epub 2019 Jul 20. PMID 31327102
- [Background] Morisson L, Nadeau-Vallee M, Espitalier F, Laferriere-Langlois P, Idrissi M, Lahrichi N, Gelinas C, Verdonck O, Richebe P. Prediction of acute postoperative pain based on intraoperative nociception level (NOL) index values: the impact of machine learning-based analysis. J Clin Monit Comput. 2023 Feb;37(1):337-344. doi: 10.1007/s10877-022-00897-z. Epub 2022 Aug 4. PMID 35925430
- [Background] Neumann C, Gehlen L, Weinhold L, Strassberger-Nerschbach N, Soehle M, Kornilov E, Thudium M. Influence of Intraoperative Nociception during Hip or Knee Arthroplasty with Supplementary Regional Anaesthesia on Postoperative Pain and Opioid Consumption. Medicina (Kaunas). 2023 Jun 17;59(6):1166. doi: 10.3390/medicina59061166. PMID 37374370
- [Result] Gelinas C, Shahiri T S, Richard-Lalonde M, Laporta D, Morin JF, Boitor M, Ferland CE, Bourgault P, Richebe P. Exploration of a Multi-Parameter Technology for Pain Assessment in Postoperative Patients After Cardiac Surgery in the Intensive Care Unit: The Nociception Level Index (NOL)TM. J Pain Res. 2021 Dec 7;14:3723-3731. doi: 10.2147/JPR.S332845. eCollection 2021. PMID 34908872
- [Result] Shahiri TS, Richebe P, Richard-Lalonde M, Gelinas C. Description of the validity of the Analgesia Nociception Index (ANI) and Nociception Level Index (NOL) for nociception assessment in anesthetized patients undergoing surgery: a systematized review. J Clin Monit Comput. 2022 Jun;36(3):623-635. doi: 10.1007/s10877-021-00772-3. Epub 2021 Nov 16. PMID 34783941
- [Result] Ghiyasinasab M, Morisson L, Laferriere-Langlois P, Geraldo-Demers MA, Gelinas C, Nadeau-Vallee M, Verdonck O, Lahrichi N, Richebe P. Identification of the intraoperative antinociceptive effect of intravenous fentanyl using the Nociception Level (NOL) index versus clinical parameters in patients undergoing gynecological laparoscopic surgery: A secondary analysis of the NOLGYN study. Anaesth Crit Care Pain Med. 2022 Aug;41(4):101102. doi: 10.1016/j.accpm.2022.101102. Epub 2022 May 25. PMID 35643392
- [Result] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Result] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633
- [Result] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185